CLINICAL TRIAL: NCT01471080
Title: A Prospective Controlled Study on Treatment of Giant Cavernous Hemangiomas of the Liver：RFA Versus Laparoscopic Hepatectomy.
Brief Title: A Prospective Controlled Study on Treatment of Giant Cavernous Hemangiomas of the Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, feng xiaobin, Institute of hepatobiliary surgery,southwest hospital, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: swhb004
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2012-11

CONDITIONS: Laparoscopic Hepatectomy; Radio-frequency Ablation; Giant Cavernous Hemangiomas; Liver
Keywords: laparoscopic hepatectomy; radio-frequency ablation; giant cavernous hemangiomas; liver
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA group (Experimental): using RFA to treat cavernous hemangiomas
  Interventions: Procedure: RFA
- hepatectomy group (Active Comparator): using laparoscopic hepatectomy to treat cavernous hemangiomas of the liver
  Interventions: Procedure: hepatectomy

INTERVENTIONS:
Procedure: RFA — using RFA to treat cavernous hemangiomas
  Other Names: radiofrequence ablation
  Arms: RFA group
Procedure: hepatectomy — using hepatectomy to treat cavernous hemangiomas
  Other Names: liver resection
  Arms: hepatectomy group

SUMMARY:
In the past, the investigators often treated giant cavernous hemangiomas of the liver by hepatectomy.Recently RFA and laparoscopic hepatectomy are also available and could be applied to cure this disease.But we can't get a clear answer about their effectiveness and safety. Hence the investigators conduct this study to explore the effectiveness and efficiency of the these two methods and compare their short to mid-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* giant cavernous hemangiomas with a diameter larger than or equal to 5 cm diagnosed by more than one imaging modalities
* age between 18 years to 65 years
* without gender restriction
* PLT account more than 50 e9
* without abnormal of liver function test
* with substantial evidence of growing size than before
* symptom associated cavernous hemangiomas
* with a strong desire of the patients for the treatment

Exclusion Criteria:

* pregnant women
* abnormal of liver function or coagulation dysfunction and/or concurrent with sever cardiac or pulmonary disorders
* patient with a poor condition that can't bear the approach of either RFA or laparoscopic hepatectomy
* tumor size more than 20cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
disappearance rate of disease | 1 month
  to determine the disappearance rate of disease by imaging modality using enhanced Ultrasound examine and/or enhanced CT

SECONDARY OUTCOMES:
complication rate | 1 month
  obvious complications including bleeding, bile leakage will be take into account.recover rate. symptom relief and satisfactory of the treatment
hospital stay and relating overall cost for treatment | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of hepatobiliary surgery,southwest hospital, Chongqing, Chongqing Municipality, China